CLINICAL TRIAL: NCT06841263
Title: Multi-methods Study on Inclusive Cancer Diagnosis in People with Disabilities and Health Outcomes
Acronym: MICaDO
Status: Not yet recruiting | Type: Observational
Sponsor: Cristina Renzi (Other)
Collaborators: Politecnico di Milano (Other); University College, London (Other); Accademia Lombarda di Sanità Pubblica (Unknown); DAMA (Disabled Advanced Medical Assistance) (Unknown); LEDHA (League for the Rights of People with Disabilities and the Promotion of Autonomy) (Unknown); HPA (Health Protection Agency) of the Metropolitan City of Milan (Unknown)
Responsible Party: Sponsor-Investigator, Cristina Renzi, Associate Professor and Medical Doctor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: CET 470-2024; 2024-1740 (Other Grant/Funding Number: Fondazione Cariplo)
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Disabled Persons; Cancer Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Peoplewith psychiatric, intellectual, neurological, sensory and physical disabilities
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable - observational study

SUMMARY:
The MICaDO study is a multi-method study that aims to investigate inclusive cancer diagnosis in people with disabilities and health outcomes. The main objective is to examine variations in cancer diagnosis and outcomes among individuals with psychiatric, intellectual, neurological, and sensory disabilities to develop interventions aimed at improving cancer care. The hypothesis that investigators will investigate is that people with disability are diagnosed with cancer later than people without disability due to a range of barriers, including physical, sensory, cognitive, and social barriers. The study will use a mixed-methods approach, combining quantitative research (electronic health record analysis) and qualitative research (interviews). The total duration of the study is two years.

ELIGIBILITY:
Inclusion Criteria:

Electronic health record study:

* Patients with psychiatric, intellectual, neurological, and sensory disabilities who received care at San Raffaele Hospital of Milan between 2011 and 2024
* Patients without disabilities who received care at San Raffaele Hospital of Milan between 2011 and 2024 (ratio 4:1 of patients without vs. with disabilities)
* Patients with psychiatric, intellectual, neurological, and sensory disabilities recorded in the Lombardy Regional Data Warehouse between 2011 and 2024
* Patients without disabilities recorded in the Lombardy Regional Data Warehouse between 2011 and 2024 (ratio 4:1 of patients without vs. with disabilities)
* Patients aged 18 and over

Qualitative Interviews:

* Patients aged 18 and over with psychiatric, intellectual, neurological, and sensory disabilities who received care at San Raffaele Hospital of Milan, DAMA (Disabled Advanced Medical Assistance) in Territorial Social Health Companies "Santi Paolo e Carlo" and LEDHA (League for the Rights of People with Disabilities and the Promotion of Autonomy) and their caregivers
* Healthcare provider working at San Raffaele Hospital of Milan, DAMA (Disabled Advanced Medical Assistance) in Territorial Social Health Companies "Santi Paolo e Carlo" and general practitioners

Exclusion Criteria:

* Patients under 18 years of age
* Patients don't speak the Italian language (for the qualitative study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified through various sources, including inpatient hospital settings and outpatient clinics. Eligible participants will be approached and invited to participate in the study. A screening process will be conducted to evaluate eligibility based on predefined criteria. Once eligibility is confirmed, participants will be registered for the study and provided with detailed information about the procedures and their rights.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic pathways and oncological outcomes in Patients with Disabilities: | Baseline
  For the quantitative part of the study, the investigators will examine several outcomes, each measured separately comparing patients with and without specific disabilities: emergency presentation measured as a binary variable (No/Yes); diagnosis through screening measured as a binary variable (No/Yes); cancer stage at diagnosis measured as an ordinal categorical variable (Stage 1, 2, 3, 4); short-term mortality measured as a percentage rate at 30 days and 90 days from diagnosis. The data will be extracted from electronic health records at San Raffaele Hospital in Milan and the Lombardy Regional Data Warehouse.
  For the qualitative part of the study, the investigators will perform qualitative interviews with patients/caregivers and healthcare providers from the Lombardy Region. Patients with various types of disabilities will be recruited at the San Raffaele Hospital in Milan and through outreach activities by LEDHA and DAMA.

SECONDARY OUTCOMES:
Accessibility and inclusiveness in Diagnostic Services: Validation of the DfA A.U.D.I.T. | Baseline
  The investigators will employ the Design for All (DfA) A.U.D.I.T., a digital platform developed by the Design and Health Lab of the Politecnico di Milano, to examine building performance, focusing on screening and diagnostic services. Specifically, the investigators will evaluate the interaction between physical, sensory, cognitive, and social barriers to validate a DfA tool for improving accessibility, inclusivity, and equity.